CLINICAL TRIAL: NCT00846651
Title: Comparison of Phenylephrine Infusion With Colloids vs. Crystalloids for Reduction of Spinal-induced Hypotension During Cesarean Section
Brief Title: Spinal Anesthesia Induced Hypotension During Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sonia Vaida, M.D, Vice chair for research, Anesthesia Department, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #29595
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Hypotension
Keywords: spinal anesthesia; cesarean section
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- colloid, then phenylephrine infusion (Experimental): colloid administration; with 0.5 L Hydroxyethylstarch solution at a rate of 17 ml/min and completed over 30 min. A phenylephrine infusion will be started immediately after performing the spinal anesthesia and continued until time of uterine incision.
  Interventions: Other: Colloid administration; Drug: phenylephrine infusion
- crystalloid, then phenylephrine infusion (Active Comparator): crystalloid administration; The patients received 1.5 L Ringer's lactate infusion at a rate of 50 ml/min and completed over 30 min prior to spinal anesthesia for cesarean section. A phenylephrine infusion will be started immediately after performing the spinal anesthesia and continued until time of uterine incision.
  Interventions: Other: Crystalloid administration; Drug: phenylephrine infusion

INTERVENTIONS:
Other: Colloid administration — The patients received 0.5 L colloid solution (hydroxyethylstarch 6%) or 1.5 L Ringer lactate prior to spinal anesthesia for cesarean section.
  Arms: colloid, then phenylephrine infusion
Other: Crystalloid administration — The patients received 1.5 L Ringer lactate prior to spinal anesthesia for cesarean section.
  Arms: crystalloid, then phenylephrine infusion
Drug: phenylephrine infusion — A phenylephrine infusion will be started immediately after performing the spinal anesthesia and continued until time of uterine incision.

SUMMARY:
The purpose of this study is to compare two methods for preventing low blood pressure associated with spinal anesthesia during Cesarean sections.

DETAILED DESCRIPTION:
Many women experience low blood pressure after spinal anesthesia for Cesarean section. This low blood pressure may result in nausea, vomiting dizziness and impairment of uterine blood flow.The purpose of this study is to compare two methods for preventing low blood pressure associated with spinal anesthesia during Cesarean sections. In both methods, we will attempt to prevent low blood pressure using phenylephrine infusion that has been shown to be effective in recent research. In addition to receiving phenylephrine one group of patients will receive standard salt solution (Ringer's lactate solution), while the other group will receive a different, intravenous fluid called hydroxyethylstarch.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II
* Elective cesarean section
* Weight 50-120 kg, Height 150-180 cm
* Normal singleton pregnancy
* Beyond 36 weeks gestation
* No known fetal abnormalities
* Ages 18-35

Exclusion Criteria:

* Contraindications to spinal anesthesia
* Multiple gestation, placenta previa, accreta
* Pregnancy induced hypertension or preeclampsia
* Diabetes mellitus, cardiovascular diseases
* Coagulopathy
* Spinal cord abnormalities, spinal surgery, or preexisting neurological dysfunction
* Baseline HR <65
* Failed spinal anesthesia/inadequate sensory block for surgery
* History of abnormal bleeding
* History of adverse reactions to hydroxyethylstarch

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PennState Hershey Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We applied for an IRB approval for 90 patients. The power analysis indicated that a minimum of 37 subjects for each group was needed. To allow for potential dropouts, we applied for 45 patient in each group. (total of 9O patients)
Groups:
- Colloid, Then Phenylephrine Infusion: colloid administration; with 0.5 L Hydroxyethylstarch solution at a rate of 17 ml/min and completed over 30 min.A phenylephrine infusion will be started immediately after performing the spinal anesthesia and continued until time of uterine incision.
- Crystalloid, Then Phenylephrine Infusion: Crystalloid administration; 1.5 L Ringer's lactate infusion at a rate of 50 ml/min and completed over 30 min. A phenylephrine infusion will be started immediately after performing the spinal anesthesia and continued until time of uterine incision.
Period: Overall Study
Arm/Group | Colloid, Then Phenylephrine Infusion | Crystalloid, Then Phenylephrine Infusion
Started | 41 | 41
Completed | 37 | 37
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colloid, Then Phenylephrine Infusion | Crystalloid, Then Phenylephrine Infusion | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 41 | 82
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (5.1) | 28.3 (5.9) | 26.6 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 82
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 41 | 82

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Maternal Hypotension
Time Frame: participants were assessed for an average of 20 min, after performing the spinal anesthetic till the delivery of the baby
Measure: Number; unit: percentage of participants
Arm/Group | Colloid, Then Phenylephrine Infusion | Crystalloid, Then Phenylephrine Infusion
Number analyzed (Participants) | 37 | 37
percentage of participants | 10.8 | 27

2. Secondary Outcome: Dosage of Phenylephrine Used
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg of phenylephrine
Arm/Group | Colloid, Then Phenylephrine Infusion | Crystalloid, Then Phenylephrine Infusion
Number analyzed (Participants) | 37 | 37
mcg of phenylephrine | 1077 (541) | 1477 (591)

3. Secondary Outcome: Incidence of Maternal Bradycardia
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Colloid, Then Phenylephrine Infusion | Crystalloid, Then Phenylephrine Infusion
Number analyzed (Participants) | 37 | 37
percentage of participants | 35.1 | 45.8

4. Secondary Outcome: Fetal Cord Blood pH
Time Frame: delivery of the baby
Population: Physician policy changes resulted in blood gas values not being ordered and thus data was not available for the outcome measure.
Arm/Group | Colloid, Then Phenylephrine Infusion | Crystalloid, Then Phenylephrine Infusion
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: APGAR Scores
Description: The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10 with higher scores being better than lower scores. The five criteria are summarized using words chosen to form an acronym (Appearance, Pulse, Grimace, Activity, Respiration).
Time Frame: Apgar scores were assessed at 1 amd 5 min after delivery of the baby
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Colloid, Then Phenylephrine Infusion | Crystalloid, Then Phenylephrine Infusion
Number analyzed (Participants) | 37 | 37
units on a scale | 9 [7 to 10] | 9 [8 to 10]

6. Secondary Outcome: Incidence of Maternal Nausea and Vomiting
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Colloid, Then Phenylephrine Infusion | Crystalloid, Then Phenylephrine Infusion
Number analyzed (Participants) | 37 | 37
percentage of participants | 16.2 | 18.9

ADVERSE EVENTS:
Arm/Group | Colloid, Then Phenylephrine Infusion | Crystalloid, Then Phenylephrine Infusion
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

LIMITATIONS AND CAVEATS:
technical problems for analysing fetal pH in all newborns

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No